CLINICAL TRIAL: NCT05171426
Title: Incidental Cancer in Colectomy Specimens From Patients With Familial Adenomatous Polyposis
Brief Title: Incidental Cancer in Familial Adenomatous Polyposis
Status: Completed | Type: Observational
Sponsor: Dr. Ersin Arslan Education and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Uylas, Primary investigator, Tepecik Training and Research Hospital
Other Study IDs: 2018/16-20
Record Dates: First submitted 2021-12-10; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Cancer
Keywords: familial adenomatous polyposis; colectomy; rectum; cancer; adenoma
MeSH Terms: conditions — Neoplasms; Adenomatous Polyposis Coli; Adenoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- incidental cancer: familial adenomatous polyposis with incidental cancer

SUMMARY:
Colectomy is life-saving in patients with familial adenomatous polyposis (FAP) because cancer development is inevitable in individuals with this disease. In this study, we aimed to determine the incidence of incidental malignancy in surgical specimens from patients who underwent colectomy for FAP. Prophylactic colectomy should be performed in patients with FAP, as colorectal cancer transformation is inevitable in these individuals. The possibility of incidental cancer identified via histopathological analysis of colectomy specimens should be kept in mind in these patients.

DETAILED DESCRIPTION:
Colectomy is life-saving in patients with familial adenomatous polyposis (FAP) because cancer development is inevitable in individuals with this disease. In this study, we aimed to determine the incidence of incidental malignancy in surgical specimens from patients who underwent colectomy for FAP. The files of patients diagnosed with FAP who underwent surgery in our clinic between 2010 and 2020 were retrospectively reviewed. Definitive surgery was performed in patients with histopathological malignancy identified in colonoscopic biopsies in the preoperative period, while prophylactic surgery was performed in patients without malignancy. The incidence of incidental malignancy in histopathological specimens from patients who underwent prophylactic colectomy was determined. Prophylactic colectomy should be performed in patients with FAP, as colorectal cancer transformation is inevitable in these individuals. The possibility of incidental cancer identified via histopathological analysis of colectomy specimens should be kept in mind in these patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Familial Adenomatous Polyposis

Exclusion Criteria:

* did not receive surgical treatment
* data deficiencies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Familial Adenomatous Polyposis patients
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
incidental cancer | 2 or 3 week
  Familial Adenomatous Polyposis with cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Ersin Arslan Training and Resource Hospital, Gaziantep, Turkey (Türkiye)